CLINICAL TRIAL: NCT06216587
Title: A Randomized, Double-blind Controlled Trial to Assess the Impact of BLa80 on the Intestinal Health of Individuals Who Consume Alcohol
Brief Title: BLa80 Improve Drinkers' Gut Microbiota
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2023008
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Alcohol Drinking, Adult Disease
MeSH Terms: conditions — Alcohol Drinking; Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: BLa80
- Probiotic group (Experimental)
  Interventions: Dietary Supplement: BLa80

INTERVENTIONS:
Dietary Supplement: BLa80 — Collect patient fecal samples, test for 16S rRNA, and analyze the changes in the patient's gut microbiota before and after taking BLa80.

SUMMARY:
The goal of this clinical trial is to understand the effects of the probiotic BLa80 on the gut health of people who drink alcohol regularly. We want to find out if this probiotic can help improve the health of the digestive system in those who consume alcohol. The main questions we aim to answer are: Does BLa80 positively change the composition of gut bacteria in alcohol consumers? Participants in this study will: Be randomly assigned to one of two groups. One group will receive the probiotic BLa80, and the other group will receive a placebo (a substance with no active therapeutic effect). Take their assigned treatment for a specified period, as directed by the study protocol. Undergo regular health checks and provide feceal samples for analysis to see how their gut bacteria might have changed during the study. This study is important because it explores whether a specific type of probiotic can help protect or improve gut health in people who drink alcohol, potentially offering a new way to support digestive health.

ELIGIBILITY:
Inclusion Criteria:

Aged 19-45 years, currently consuming alcohol (defined as having consumed alcohol on at least one day in the past 30 days); Willing to voluntarily agree to and comply with the trial protocol, and capable of timely participation in screening and follow-up; No symptoms of alcohol allergy, with a history of alcohol consumption; Have not suffered from gastrointestinal diseases in the past month; Have not taken antibiotics in the past month.

Exclusion Criteria:

Individuals under 19 or over 45 years of age, with an allergic constitution or allergy to any component of the test substance, symptoms of alcohol allergy, and pregnant or breastfeeding women; Those who experience discomfort such as diarrhea or bloating after taking the test substance; Patients with serious diseases of the cardiovascular, liver, kidney, hematopoietic systems, autoimmune diseases, endocrine disorders, mental illnesses, existing high blood sugar, or unhealthy gastrointestinal conditions; Those who discontinue the test sample or take other medications midway, making it difficult to judge efficacy or with incomplete data; Recently taken probiotics, prebiotics, or antibiotics related to the function of the test substance, affecting the judgment of results; Individuals with a daily diet that is either too light or too greasy; those with special dietary structures due to weight loss or other reasons (such as a ketogenic diet); Individuals with low body fat, BMI < 23.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-06-25 (Estimated); Study Completion 2024-07-14 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiota | 8 weeks
  Collect patient fecal samples, test for 16S rRNA